CLINICAL TRIAL: NCT00890214
Title: Heparin Versus Prostacyclin in Continuous Hemodiafiltration for Acute Renal Failure: Effects on Platelet Responsiveness in the Systemic Circulation and Across the Filter.
Brief Title: Prostacyclin's Effect on Platelet Responsiveness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Massimo Antonelli, Istituto di Anestesia e Rianimazione
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AABR-0609
Record Dates: First submitted 2009-04-23; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Acute Kidney Failure
Keywords: Anticoagulation; Prostacyclin; Heparin; Renal Replacement Therapy; Kidney failure acute; Platelet aggregation
MeSH Terms: conditions — Acute Kidney Injury | interventions — Epoprostenol; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 prostacyclin group (Active Comparator): prostacyclin analogue (PGIA) used as circuit anticoagulant during continuous venovenous hemodiafiltration (CVVHDF) in acute kidney failure patients
  Interventions: Drug: prostacyclin
- 2 heparin group (Active Comparator): unfractionated heparin used as circuit anticoagulant during continuous venovenous hemodiafiltration (CVVHDF) in acute kidney failure patients
  Interventions: Drug: heparin

INTERVENTIONS:
Drug: prostacyclin — prostacyclin was infused as CRRT circuit anticoagulant into the arterial-line of the circuit at 4 ng/Kg/min
  Other Names: prostacyclin epoprostenol (PGIA) (Flolan®, Glaxo-Wellcome)
  Arms: 1 prostacyclin group
Drug: heparin — was prepared using our standard protocol: 2 ml of an already-stored solution containing 5000 IU/ml of UFH were diluted in 20 ml of saline obtaining a final concentration of 500 IU/ml, and infused pre-filter at 6 IU/Kg/h, according to the post-filter activated clotting time measured hourly, and adjusted to obtain a value between 180 and 200 sec.
  Other Names: unfractionated heparin UFH (Liquemin®, Roche).
  Arms: 2 heparin group

SUMMARY:
The researchers investigated the influence of a prostacyclin analogue (PGIA) versus unfractionated heparin (UFH) on ex vivo platelet function, during continuous venovenous hemodiafiltration.

DETAILED DESCRIPTION:
Context and purpose of the study: Prospective, randomized comparison of a PGIA versus UFH as circuit anticoagulant. Platelet responsiveness was assessed from peripheral blood by light-transmittance aggregometry (LTA) induced by collagen and ADP, at baseline, 4 and 24 hrs after treatment onset. Platelet function was also assessed in blood samples collected in the circuit before and after the filter. The Setting was a University Hospital Intensive Care Unit. 23 ICU patients with Acute Renal Failure needing CVVHDF were studied during standard CVVHDF therapy, at random infusion in the extracorporeal circuit of PGIA or UFH.

ELIGIBILITY:
Inclusion Criteria:

* critically patients ill patients with acute kidney failure (AKI) needing renal replacement therapy

Exclusion Criteria:

* therapy with aspirin or other non-steroidal anti-inflammatory drugs in the previous 7 days
* concomitant treatment with other extracorporeal organ-assist devices any other drug affecting coagulation or platelets

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, MD, Study Director — Istituto Anestesia e Rianimazione Università Cattolica Policlinico Gemelli
Locations (1):
- Policlinico Gemelli, Rome, Italy

REFERENCES:
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078